CLINICAL TRIAL: NCT07086664
Title: An Interventional Phase 1b, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study to Investigate the Safety, Tolerability, and Pharmacodynamic Effect of PF-07258669 Compared to Placebo in Older Participants Including Those at Risk of Malnutrition
Brief Title: A Study to Learn About the Study Medicine Called PF-07258669 in Older Adults Including Those at Risk of Malnutrition
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely discontinued due to a business decision. The decision to terminate the study is not related to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C4541011; 2025-520763-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: Malnutrition risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-07258669 (Experimental)
  Interventions: Drug: PF-07258669

INTERVENTIONS:
Drug: Placebo — Oral tablet
  Arms: Placebo
Drug: PF-07258669 — Oral tablet
  Arms: PF-07258669

SUMMARY:
The purpose of this study is to look at safety, tolerability, and pharmacodynamic effects (i.e. how the study drug affects your body) of PF-07258669 in older participants ((60 years to <90 years) including those at risk of malnutrition.

The study medicine PF-07258669 is being developed for the treatment of unintended weight loss in older adults. People with this condition have decreased appetite and food intake, which is an important reason for poor nutrition and health results in people with unintended weight loss.

This is approximately a 26-week-long study with 9 visits to the study doctor and 4 telehealth visits (ie. visits by phone call). The study will include

* Screening period for up to 4 weeks
* Pre-treatment period of 2 weeks
* Treatment period of 16 weeks : study drug (PF-07258669 or matching placebo)
* Follow-up period of 4 weeks The study requires answering questionnaires and use of digital devices at home to measure blood pressure and physical activity. The study team will monitor how each participant is doing during the study

ELIGIBILITY:
Inclusion Criteria Are 60 years to <90 years Are males or females who can no longer have children Have Body weight ≥40 kg and Body mass index (BMI) ≤25 kg/m2 Exclusion Criteria Evidence or history of clinically significant medical conditions. Positive for active, untreated HIV, hepatitis B, and/or hepatitis C History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.

Voluntary diet restriction or eating disorder

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events | Baseline to Week 20

SECONDARY OUTCOMES:
Percent change from baseline in body weight | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (10):
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - JEM Research Institute, Atlantis, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - De La Cruz Research Center, LLC, Miami, Florida
  - Headlands Research Orlando, Orlando, Florida
  - AA Medical Research Center, Flint, Michigan
  - Clinical Research Professionals, Chesterfield, Missouri
  - Javara - Nevada Health Centers - Carson City, Carson City, Nevada
  - Circuit Clinical, Secaucus, New Jersey
  - Circuit Clinical /North Hudson Community Action Corporation, West New York, New Jersey
- Canada (3):
  - Alpha Recherche Clinique, Québec, Quebec
  - Diex Recherche Inc. Division Victoriaville, Victoriaville, Quebec
  - Centre de Recherche Saint-Louis inc., Québec
- Yao Tokushukai General Hospital, Yao Shi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4541011